CLINICAL TRIAL: NCT06684132
Title: Effects of Respiratory Muscle Training in Patients With Scleroderma With Pulmonary Involvement
Brief Title: Respiratory Muscle Training in Scleroderma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/13-06
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Scleroderma (Limited and Diffuse)
Keywords: Scleroderma; Inspiratory muscle training; pulmonary functions
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): High intensity intermittent inspiratory muscle training (H-IMT) will be applied. This training will be performed with Power breath (POWERbreathe Classic Light Resistance, PowerBreath, IMT Technologies Ltd, Birmingham, UK) respiratory muscle training device. The H-IMT will be performed in seven sets of three-minute cycles consisting of two minutes of training followed by one minute of rest in the training workload. Each session will consist of 14 minutes of loading and seven minutes of rest for a total of 21 minutes.
  Interventions: Other: Inspiratory muscle training
- Exercise group (Other): Stretching exercises for pectoral muscles, neck muscles and back muscles, strengthening exercises for upper extremity and back muscles and posture exercises will be applied.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Inspiratory muscle training — The H-IMT will be performed in seven sets of three-minute cycles consisting of two minutes of training followed by one minute of rest in the training workload. Each session will consist of 14 minutes of loading and seven minutes of rest for a total of 21 minutes.
  Arms: IMT group
Other: Exercise — Stretching exercises for pectoral muscles, neck muscles and back muscles, strengthening exercises for upper extremity and back muscles and posture exercises will be applied.
  Arms: Exercise group

SUMMARY:
The aim of this study is to investigate the effects of IMT on respiratory muscle strength, pulmonary function tests, quality of life aerobic capacity, dyspnea, fatigue and physical activity level in scleroderma patients with ILD. The study will include 30 Scleroderma + ILD patients who are under follow-up in Fırat University Rheumatology Department. Patients will be randomly divided into two groups. High intensity intermittent inspiratory muscle training (H-IMT) will be applied to the respiratory muscle training group in addition to the exercise program. Respiratory muscle strength will be assessed by maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP); aerobic capacity will be assessed by exercise test and VO2max. Dyspnea will be assessed with the Modified Medical Research Council Scale; fatigue with the Fatigue Severity Scale; quality of life with the Scleroderma Health Assessment Questionnaire; physical activity level with the International Physical Activity Scale - Short Form

DETAILED DESCRIPTION:
Inspiratory muscle training (IMT) is performed by inspiring against an external load provided by a device. It is easy to implement, low cost and can be easily integrated into rehabilitation programs. Pulmonary rehabilitation and inspiratory muscle training have been applied as an effective method in ILD. However, there are no studies investigating the effects of IMT in individuals with ILD. The aim of this study was to investigate the effects of IMT on respiratory muscle strength, pulmonary function tests, quality of life, aerobic capacity, dyspnea, fatigue and physical activity level in scleroderma patients with ILD. The study will include 30 Scleroderma + ILD patients who are under follow-up in Fırat University Rheumatology Department. Patients will be randomly divided into two groups. High intensity intermittent inspiratory muscle training (H-IMT) will be applied to the respiratory muscle training group in addition to the exercise program. This training will be performed with Power breath (POWERbreathe Classic Light Resistance, PowerBreath, IMT Technologies Ltd, Birmingham, UK) respiratory muscle training device. In the control group, only stretching, strengthening and posture exercises will be applied as a home program. Respiratory muscle strength will be assessed by maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP); aerobic capacity will be assessed by VO2max with exercise test. dyspnea will be assessed using the Modified Medical Research Council Scale; fatigue will be assessed using the Fatigue Severity Scale; quality of life will be assessed using the Scleroderma Health Assessment Questionnaire; physical activity level will be assessed using the International Physical Activity Scale - Short Form.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Patients whose medical treatment has not changed in the last three months
* Patients who volunteered to participate in the study and were cooperative
* Literate patients
* Patients followed with a diagnosis of SSc

Exclusion Criteria:

* Patients who are pregnant
* Patients with a diagnosis of malignancy
* Patients with other concomitant systemic inflammatory rheumatic diseases
* Patients with neurological, orthopedic or congenital problems that prevent physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | up to 8 weeks
  Respiratory muscle strength will be assessed with an intraoral pressure gauge. Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) are commonly used non-invasive methods to determine respiratory muscle strength. These are intraoral pressures measured at maximum respiration against a valve that closes the airways. When applying MIP, the patient is asked to perform maximal expiration.

SECONDARY OUTCOMES:
Fatigue | up to 8 weeks
  Fatigue will be assessed with the Fatigue Severity Scale (FSS), the Turkish validity and reliability of which was performed by Armutlu et al.